CLINICAL TRIAL: NCT06599723
Title: Racz Catheter Technique Versus Conventional Technique in Lumbar Epidural Steroid Injection for Management of Low Back Pain: A Randomized Controlled Trial
Brief Title: Racz Catheter Technique Versus Conventional Technique in Lumbar Epidural Steroid Injection for Management of Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR800/8/24
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Racz Catheter; Conventional; Lumbar; Epidural; Steroid Injection; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional lumbar steroid injections group (Active Comparator): Patients will receive conventional lumbar steroid injections.
  Interventions: Drug: Conventional lumbar steroid injections
- Racz catheter group (Experimental): Patients will receive lumbar epidural steroid using Racz catheter.
  Interventions: Procedure: Racz catheter

INTERVENTIONS:
Drug: Conventional lumbar steroid injections — Patients will receive conventional lumbar steroid injections.
  Arms: Conventional lumbar steroid injections group
Procedure: Racz catheter — Patients will receive lumbar epidural steroid using Racz catheter.
  Arms: Racz catheter group

SUMMARY:
The aim of this study is to compare Racz catheter technique and conventional technique in lumbar epidural steroid injection for the management of low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is defined as a localized discomfort sensation below the costal margin and above the inferior gluteal folds, with or without leg pain. Conservative treatment for LBP is focused on delaying or preventing the need for surgery. Indeed, LBP can improve spontaneously or with non-surgical treatment. However, cases that fail to improve with conservative management may need to be considered for a surgical approach.

The epidural injection is a well-founded anesthetic and analgesic technique; moreover, nowadays, new technological devices can help anesthesiologists to learn and to administer it. One of these devices is Racz catheter epidural adhesiolysis. Racz catheter epidural adhesiolysis treatment addresses two issues, the injectate always reaches the area being targeted also the injections are likely to loosen fibrotic adhesions which may be the main cause of the pain in some cases.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* Patients suffering from persistent lumbar pain, grade 1 spondylolisthesis, facet osteoarthropathy, and small disc on radiological findings.

Exclusion Criteria:

* Uncooperative patients.
* Contraindications to perform the proper technique e.g., coagulopathy and skin infection.
* History of allergy to contrast medium.
* Rupture disc.
* Lumbar canal stenosis.
* Previously operated traditional spine surgeries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Oswestry score | 6 month post-procedure
  Oswestry Low Back Disability Questionnaire: This questionnaire has been designed to give us information as to how back pain has affected a patient's ability to manage everyday life. It consists of 10 questions for each question, there is a possible 5 points (0 for the first answer, 1 for the second answer, etc). Add up the total for the 10 questions and rate them on the scale (0-4 no disability, 5-14 mild disability, 15-24 moderate disability, 25-34 severe disability, 35-50 complete disability). It will be assisted pre-procedure as a baseline, after 1, 2, 4, 6 month post-procedure.

SECONDARY OUTCOMES:
Degree of pain | 6 month post-procedure
  The degree of pain will be assessed using the visual analog scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable").
Patient satisfaction | 6 month post-procedure
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Procedure technique time | Intraoperatively
  The time consumed to perform both techniques will be recorded.
Incidence of complications | 6 month post-procedure
  Complications that may occur during the technique such as (bending of the tip of the needle, shearing of the catheter, misplacement of the catheter, blocking of the catheter, blood aspiration and bleeding in the epidural space, hypotension, migration of the catheter, paresthesia, headache and infection) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author